CLINICAL TRIAL: NCT02653092
Title: Reprometabolic Syndrome Mediates Subfertility in Obesity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-1052; UL1TR001082 (NIH)
Record Dates: First submitted 2016-01-05; First posted 2016-01-12 (Estimated); Results first posted 2023-06-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Infertility; Hypogonadotropic Hypogonadotropism; Hyperinsulinemia
MeSH Terms: conditions — Obesity; Infertility; Hyperinsulinism | interventions — Insulin; Insulin, Regular, Human; soybean oil, phospholipid emulsion; Fatty Acids, Nonesterified; Glucose; Heparin; Anticoagulants; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aim 1-Administration of FFA in an acute model (Active Comparator): Reproduction of the reproductive phenotype of obesity in Normal Weight Women (NWW) by:
  1) infusing insulin and free fatty acids (FFAs) in short term experiments and measuring gonadotropin pulsatility and pituitary GnRH response Assessment of the gluco-regulatory and anti-lipolytic actions of insulin with a 2-stage, Hyperinsulinemic, Euglycemic Clamp (HEC) to evaluate both suppression of lipolysis and hepatic glucose production.
  Interventions: Drug: Insulin; Drug: Intralipid; Drug: Dextrose; Drug: Heparin; Drug: GnRH
- Aim 2-Hyperinsulinemic Euglycemic Clamp after a chronic administration of a diet (Experimental): Assessment of the gluco-regulatory and anti-lipolytic actions of insulin with a 2-stage, Hyperinsulinemic, Euglycemic Clamp (HEC) to evaluate both suppression of lipolysis and hepatic glucose production.
  Inducing a chronic model of the reprometabolic syndrome by administering a eucaloric diet that is relatively high in pro-inflammatory omega-6 fatty acids and low in anti-inflammatory omega-3 fatty acids (high fat diet; HFD) for one month while monitoring gonadotropin pulsatility and daily urinary reproductive hormone excretion.
  Interventions: Drug: Insulin; Drug: Dextrose; Drug: Heparin; Drug: GnRH; Procedure: Hyperinsulinemic Euglycemic Clamp

INTERVENTIONS:
Drug: Insulin
  Other Names: Humulin
Drug: Intralipid
  Other Names: Free Fatty Acid
  Arms: Aim 1-Administration of FFA in an acute model
Drug: Dextrose
  Other Names: d-glucose
Drug: Heparin
  Other Names: anticoagulant
Drug: GnRH
  Other Names: gonadorelin acetate
Procedure: Hyperinsulinemic Euglycemic Clamp
  Other Names: HEC
  Arms: Aim 2-Hyperinsulinemic Euglycemic Clamp after a chronic administration of a diet

SUMMARY:
Obesity plays an adverse role at every stage of conception and pregnancy and mounting evidence implicates relative hypogonadotropic hypogonadism, and reduced menstrual cycle hormone secretion as likely contributors to the subfertility phenotype and possible contributors to complications of pregnancy and the developmental origin of adult diseases such as diabetes and cardiovascular disease. This study will be the first comprehensive investigation to tie together the patterns of hyperinsulinemia, hyperlipidemia and inflammation, characteristic of obesity and obesity-caused relative hypogonadotropic hypogonadotropism and its potential adverse reproductive outcomes. The investigators findings will be used to inform a subsequent clinical intervention to optimize reproductive outcomes for obese women and their offspring.

DETAILED DESCRIPTION:
Before any of the well-known adverse effects in pregnancy2,3, obesity causes a relatively hypogonadotropic hypogonadal phenotype. Reduced LH, FSH, estradiol (E2) and progesterone secretion are well documented during the menstrual cycles of obese women compared to normal weight women (NWW).4,5. Decreased gonadotropin secretion associated with obesity is related to reduced pituitary sensitivity to GnRH6. This reduction in pituitary sensitivity suggests mediation by circulating factors such as cytokines, insulin, or other pro-inflammatory signals known to be elevated in obesity. We have recently discovered that the combination of hyperinsulinemia and circulating free fatty acids (FFAs), but neither agent alone, can acutely decrease gonadotropin secretion in NWW as well as men, establishing a direct causal linkage for the central hypothesis of this proposal: that chronic pituitary suppression partially mediates obesity related subfertility. Our working model is that the combination of excess, possibly pro-inflammatory (omega-6) circulating FFAs and insulin resistance associated with obesity, cause decreased pituitary sensitivity to GnRH, with a resulting relative sex steroid deficit that further exacerbates the obese phenotype. We have named this phenotype the reprometabolic syndrome. We propose to examine the interrelationships among obesity, reproductive dysfunction and metabolic dysfunction in a mechanistic fashion. We will induce the hypogonadotropic hypogonadal phenotype of obesity in NWW, who will be primed with a high-fat diet (HFD) designed to increase circulating FFAs and produce short-term insulin resistance and higher insulin levels.1,7-11 Before and after priming, we will test the additive effects of lipid excess, insulin, and inflammation on the reproductive and metabolic axes.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) at least 18 but less than 25 kg/m2
* No history of chronic disease affecting hormone production, metabolism, or clearance
* No use of medications known to alter or interact with reproductive hormones or insulin metabolism (e.g. thiazolidinediones, metformin)
* No use of reproductive hormones within 3 months of enrollment
* Normal prolactin and thyroid stimulating hormone levels at screening
* History of regular menstrual cycles every 25-35 days
* Use of a reliable method of contraception (female or male partner sterilization; intra uterine device (IUD); abstinence; diaphragm)
* Normal hemoglobin A1c
* Screening hemoglobin >11gm/dl

Exclusion Criteria:

* Women with a baseline dietary assessment indicative of >35% daily calorie consumption from fat (as calculated based upon initial screening survey) will be excluded, as the impact of increasing their dietary fat intake may be minimal.
* Women with fasting triglycerides >300mg/dl at screening will be excluded, as they might be at risk for acute elevation of triglycerides and even pancreatitis if placed on a high fat diet
* Inability to comply with the protocol. Individuals who travel frequently, or who eat most of their meals outside of their home will be excluded, as it will be difficult to impossible for them to comply with the diet, to pick up the food cartons, etc.
* Because high proportions of dairy fat will be needed to attain 48% calories from fat in the diet, vegans and lactose intolerant individuals will be excluded.
* Pregnant women or women planning to become pregnant will be excluded.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2025-12-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Santoro, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen T, Kuhn K, Bolt M, Duffy K, Bradford AP, Santoro N. Analysis of Inflammatory Markers in Response to Induction of Reprometabolic Syndrome by a Eucaloric High Fat Diet in Normal Weight Women. Reprod Sci. 2024 Sep;31(9):2820-2828. doi: 10.1007/s43032-024-01586-9. Epub 2024 May 6. PMID 38710978
- [Derived] Santoro N, Schauer IE, Kuhn K, Fought AJ, Babcock-Gilbert S, Bradford AP. Gonadotropin response to insulin and lipid infusion reproduces the reprometabolic syndrome of obesity in eumenorrheic lean women: a randomized crossover trial. Fertil Steril. 2021 Aug;116(2):566-574. doi: 10.1016/j.fertnstert.2021.03.005. Epub 2021 Apr 8. PMID 33838870

RESULTS

PARTICIPANT FLOW:
Groups:
- Aim 1-Acute Infusion of FFA and Chronic Model: Reproduction of the reproductive phenotype of obesity in Normal Weight Women (NWW) by:
  1. infusing insulin and free fatty acids (FFAs) in short term experiments and measuring gonadotropin pulsatility and pituitary GnRH response; and
  2. inducing a chronic model of the reprometabolic syndrome by administering a eucaloric diet that is relatively high in pro-inflammatory omega-6 fatty acids and low in anti-inflammatory omega-3 fatty acids (high fat diet; HFD) for one month while monitoring gonadotropin pulsatility and daily urinary reproductive hormone excretion.
  Insulin
  Intralipid
  Dextrose
  Heparin
  GnRH
- Aim 2- Hyperinsulinemic Euglycemic Clamp: Assessment of the gluco-regulatory and anti-lipolytic actions of insulin with a 2-stage, Hyperinsulinemic, Euglycemic Clamp (HEC) to evaluate both suppression of lipolysis and hepatic glucose production.
  Insulin
  Intralipid
  Dextrose
  Heparin
  GnRH
  Hyperinsulinemic Euglycemic Clamp
Period: Overall Study
Arm/Group | Aim 1-Acute Infusion of FFA and Chronic Model | Aim 2- Hyperinsulinemic Euglycemic Clamp
Started | 26 | 58
Completed | 13 | 18
Not Completed | 13 | 40

BASELINE CHARACTERISTICS:
Groups:
- Aim 1: Reproduction of the reproductive phenotype of obesity in Normal Weight Women (NWW) by infusing insulin and free fatty acids (FFAs) in short term experiments and measuring gonadotropin pulsatility and pituitary GnRH response; and
  Insulin
  Intralipid
  Dextrose
  Heparin
  GnRH
- Aim 2: Assessment of the gluco-regulatory and anti-lipolytic actions of insulin with a 2-stage, Hyperinsulinemic, Euglycemic Clamp (HEC) to evaluate both suppression of lipolysis and hepatic glucose production before and after a eucaloric high-fat diet. Reproduction of the reproductive phenotype of obesity in Normal Weight Women (NWW) by inducing a chronic model of the reprometabolic syndrome by administering a eucaloric diet that is relatively high in pro-inflammatory omega-6 fatty acids and low in anti-inflammatory omega-3 fatty acids (high fat diet; HFD) for one month while monitoring gonadotropin pulsatility and daily urinary reproductive hormone excretion.
  Insulin
  Dextrose
  Heparin
  GnRH
  Hyperinsulinemic Euglycemic Clamp
- Total: Total of all reporting groups
Arm/Group | Aim 1 | Aim 2 | Total
Number analyzed (Participants) | 26 | 58 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 58 | 84
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.63 (5.46) | 29.53 (6.17) | 30.01 (5.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 58 | 84
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 23 | 50 | 73
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 0 | 2 | 2
  White | 21 | 44 | 65
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 26 | 58 | 84
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.60 (1.32) | 21.57 (1.97) | 21.58 (1.65)
Hormones [Count of Participants; unit: Participants] | 26 | 58 | 84

OUTCOME MEASURES:

1. Primary Outcome: Change in LH Pulse Amplitude Before and After Acute or Chronic FFA Administration
Description: LH-Luteinizing Hormone Pulse Amplitude before and after administration of FFAs. This is a measure of the post supplementation frequent blood sampling session and the baseline session.
Time Frame: First 4 hours of the frequent blood sampling study before and after FFA administration
Population: There were only 15 women who completed Aim 1 of the study. There were 19 women who completed aim 2 of the study and one had to be excluded due to not meeting the inclusion criteria once in the study.
Measure: Mean (Standard Error); unit: IU/L
Groups:
- Aim 1-Supplementation of FFAs in an Acute or Chronic Model.: Reproduction of the reproductive phenotype of obesity in Normal Weight Women (NWW) by:
  1. infusing insulin and free fatty acids (FFAs) in short term experiments and measuring gonadotropin pulsatility and pituitary GnRH response; and
  2. inducing a chronic model of the reprometabolic syndrome by administering a eucaloric diet that is relatively high in pro-inflammatory omega-6 fatty acids and low in anti-inflammatory omega-3 fatty acids (high fat diet; HFD) for one month while monitoring gonadotropin pulsatility and daily urinary reproductive hormone excretion.
  Insulin
  Intralipid
  Dextrose
  Heparin
  GnRH
- Aim 2-Hyperinsulinemic Euglycemic Clamp.: Assessment of the gluco-regulatory and anti-lipolytic actions of insulin with a 2-stage, Hyperinsulinemic, Euglycemic Clamp (HEC) to evaluate both suppression of lipolysis and hepatic glucose production.
  Insulin
  Intralipid
  Dextrose
  Heparin
  GnRH
  Hyperinsulinemic Euglycemic Clamp
Arm/Group | Aim 1-Supplementation of FFAs in an Acute or Chronic Model. | Aim 2-Hyperinsulinemic Euglycemic Clamp.
Number analyzed (Participants) | 15 | 18
IU/L | 2.33 (1.21) | 2.4 (1.1)

2. Primary Outcome: Change in Steady State Amount of Glucose Metabolized at the Set Insulin Infusion Rate Under Euglycemic Conditions
Description: Primary outcome will be M, which represents the steady state amount of glucose metabolized at the set insulin infusion rate under euglycemic conditions, which is equal to the glucose infused when the participant is euglycemic during the second stage of the HEC49. The final 30 minutes of the clamp period will be considered steady state. Glucose concentrations will be determined with the glucose oxidase method (Beckman Glucose Analyzer 2; Beckman Instruments, Fullerton, CA), while ELISA methods will be used for insulin measurements (Alpco, Salem, NH).
Time Frame: 30 minutes
Population: Aim 1 included 15 participants who completed the studies. In Aim 2 one participant was excluded due to the fact once the analysis was completed she did not meet the inclusion/exclusion criteria and the total number of participants who completed the clamp was 15 per study design.
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Aim 1-Acute and Chronic Administration of FFAs.: Reproduction of the reproductive phenotype of obesity in Normal Weight Women (NWW) by infusing insulin and free fatty acids (FFAs) in short term experiments and measuring gonadotropin pulsatility and pituitary GnRH response; and
  Insulin
  Intralipid
  Dextrose
  Heparin
  GnRH
- Aim 2-Hyperinsulinemic Euglycemic Clamp: Assessment of the gluco-regulatory and anti-lipolytic actions of insulin with a 2-stage, Hyperinsulinemic, Euglycemic Clamp (HEC) to evaluate both suppression of lipolysis and hepatic glucose production before and after a eucaloric high-fat diet. Reproduction of the reproductive phenotype of obesity in Normal Weight Women (NWW) by inducing a chronic model of the reprometabolic syndrome by administering a eucaloric diet that is relatively high in pro-inflammatory omega-6 fatty acids and low in anti-inflammatory omega-3 fatty acids (high fat diet; HFD) for one month while monitoring gonadotropin pulsatility and daily urinary reproductive hormone excretion.
  Insulin
  Dextrose
  Heparin
  GnRH
  Hyperinsulinemic Euglycemic Clamp
Arm/Group | Aim 1-Acute and Chronic Administration of FFAs. | Aim 2-Hyperinsulinemic Euglycemic Clamp
Number analyzed (Participants) | 15 | 15
mg/dL | 1.98 (0.14) | 0.0485 (0.0641)

3. Secondary Outcome: Change in GnRH Response Before and After Acute or Chronic FFA Administration
Description: GnRH response will be compared between the non-intervention and intervention study as described above for gonadotropin pulsatility. The Investigator have used area under the curve methods to determine the LH response to exogenous GnRH and will utilize the same methodology as the investigator have done in the past.
Time Frame: After the administration of GnRH at each FSS before and after acute and chronic FFA administration was assessed for up to 4 hours.
Population: All participants completed both Aim 1 and Aim 2 in the study.
Measure: Mean (Standard Error); unit: IU/L*min
Groups:
- Aim 1-Administration of FFA in an Acute Model: Reproduction of the reproductive phenotype of obesity in Normal Weight Women (NWW) by:
  1) infusing insulin and free fatty acids (FFAs) in short term experiments and measuring gonadotropin pulsatility and pituitary GnRH response Assessment of the gluco-regulatory and anti-lipolytic actions of insulin with a 2-stage, Hyperinsulinemic, Euglycemic Clamp (HEC) to evaluate both suppression of lipolysis and hepatic glucose production.
  Insulin
  Intralipid
  Dextrose
  Heparin
  GnRH
- Aim 2-Hyperinsulinemic Euglycemic Clamp After a Chronic Administration of a Diet: Assessment of the gluco-regulatory and anti-lipolytic actions of insulin with a 2-stage, Hyperinsulinemic, Euglycemic Clamp (HEC) to evaluate both suppression of lipolysis and hepatic glucose production.
  Inducing a chronic model of the reprometabolic syndrome by administering a eucaloric diet that is relatively high in pro-inflammatory omega-6 fatty acids and low in anti-inflammatory omega-3 fatty acids (high fat diet; HFD) for one month while monitoring gonadotropin pulsatility and daily urinary reproductive hormone excretion.
  Insulin
  Dextrose
  Heparin
  GnRH
  Hyperinsulinemic Euglycemic Clamp
Arm/Group | Aim 1-Administration of FFA in an Acute Model | Aim 2-Hyperinsulinemic Euglycemic Clamp After a Chronic Administration of a Diet
Number analyzed (Participants) | 15 | 15
IU/L*min | 567.63 (1.22) | 355.12 (1.23)

4. Secondary Outcome: Change in Mean FSH Parameter Before and After Acute or Chronic FFA Administration
Description: FSH parameters will be compared between the non-intervention and intervention studies for both aims as described above for gonadotropin pulsatility. The investigator will compare mean FSH, as pulsatility of FSH is less obvious than LH.
Time Frame: Before and after FFA adminstration
Population: normal weight women
Measure: Mean (Standard Error); unit: IU/L*min
Arm/Group | Aim 1-Supplementation of FFAs in an Acute or Chronic Model. | Aim 2-Hyperinsulinemic Euglycemic Clamp.
Number analyzed (Participants) | 15 | 12
IU/L*min | 242.46 (1.23) | 158.99 (1.25)

5. Secondary Outcome: Changes in Gonadotropin Pulse Frequency
Description: The investigator will compare changes in gonadotropin pulse frequency (for LH, and if we can detect distinct FSH pulses, we will compare FSH as well), mean LH and FSH and kinetics of LH, and if possible, FSH, before and after the intervention, as previously reported
Time Frame: 4 hours
Population: Normal Weight women
Measure: Mean (Standard Error); unit: IU/L
Arm/Group | Aim 1-Supplementation of FFAs in an Acute or Chronic Model. | Aim 2-Hyperinsulinemic Euglycemic Clamp.
Number analyzed (Participants) | 15 | 12
IU/L | 2.33 (1.21) | 1.49 (1.23)

6. Secondary Outcome: Urinary Hormone Profiles Before, During and After High Fat Diet Administration.
Description: Urinary hormone profiles will be assessed for the entire cycle before and two cycles after initiation of the HFD using previously described menstrual cycle parameters suitable for urinary hormone determinations. The LH peak will be determined for all cycles that demonstrate a Progesterone increment consistent with ovulation. Follicular and luteal phase lengths will be calculated, as will integrated follicular, luteal and whole cycle LH, FSH, E1c and Progesterone. The measurement is the change in value from baseline to 4 menstrual cycles (approximately 4 months) after baseline.
Time Frame: Urinary assays will be measured for 4 menstrual cycles (approximately 4 months or 115 days)
Population: Eighteen Normal weight women urinary hormones were measured during 4 menstrual cycles which was before, during and after the high fat diet administration. We looked at the change in peak LH before and after the high fat diet.
Measure: Mean (Standard Error); unit: mIU/mg Creatinine
Groups:
- Chronic Model: Reproduction of the reproductive phenotype of obesity in Normal Weight Women (NWW) by inducing a chronic model of the reprometabolic syndrome by administering a eucaloric diet that is relatively high in pro-inflammatory omega-6 fatty acids and low in anti-inflammatory omega-3 fatty acids (high fat diet; HFD) for one month while monitoring gonadotropin pulsatility and daily urinary reproductive hormone excretion.
Arm/Group | Chronic Model
Number analyzed (Participants) | 18
mIU/mg Creatinine | -10.71 (2.2)

7. Secondary Outcome: Glucose Measurements Before and After FFA Administration.
Description: Glucose will be measured by the CTRC laboratories before and after FFA administration..
Time Frame: 60 Minutes during HEC
Reporting Status: Not Posted

8. Secondary Outcome: Comparison of RBC Lipids Before and After the FFA Administration
Description: RBC lipids will also be compared, as the investigator predict that the HFD will result in increased omega-6 rich FFAs and less omega-3 FFAs
Time Frame: 30 Minutes during the HEC
Reporting Status: Not Posted

9. Secondary Outcome: DEXA Body Composition Comparison
Description: DEXA body composition will be measured before and after the intervention.
Time Frame: 5 months-before and after the interventation.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse events were collected over 6 years
Description: participants were not at risk for mortality due the nature of intervention. The participants were monitored for AEs by the investigator.
Groups:
- Aim 1: Reproduction of the reproductive phenotype of obesity in Normal Weight Women (NWW) by:
  1. infusing insulin and free fatty acids (FFAs) in short term experiments and measuring gonadotropin pulsatility and pituitary GnRH response; and
  2. inducing a chronic model of the reprometabolic syndrome by administering a eucaloric diet that is relatively high in pro-inflammatory omega-6 fatty acids and low in anti-inflammatory omega-3 fatty acids (high fat diet; HFD) for one month while monitoring gonadotropin pulsatility and daily urinary reproductive hormone excretion.
  Insulin
  Intralipid
  Dextrose
  Heparin
  GnRH
- Aim 2: Assessment of the gluco-regulatory and anti-lipolytic actions of insulin with a 2-stage, Hyperinsulinemic, Euglycemic Clamp (HEC) to evaluate both suppression of lipolysis and hepatic glucose production.
  Insulin
  Intralipid
  Dextrose
  Heparin
  GnRH
  Hyperinsulinemic Euglycemic Clamp
Arm/Group | Aim 1 | Aim 2
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/18
Other Adverse Events (participants affected / at risk) | 1/13 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aim 1 (N=13) | Aim 2 (N=18)
Headache and Nausea (Investigations) | 1 (1) | NA — One participant had a headache and experienced nausea towards the end of the infusion/frequent blood sampling session. She was removed from the infusion and give medication for the nausea and headache.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT02653092/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT02653092/ICF_001.pdf